CLINICAL TRIAL: NCT06584175
Title: Guided Internet-Delivered Cognitive Behavioural Therapy for Adults With Tinnitus in Canada: A Randomized Controlled Trial
Brief Title: Guided ICBT for Adults With Tinnitus in Canada: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123792
Record Dates: First submitted 2024-08-29; First posted 2024-09-04 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-08

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized ICBT (Experimental): Before initiation of the program, participants in the personalized ICBT group will collaboratively work with the Guide to determine which modules of the ICBT program best meet the participant's needs/goals. The ICBT program contains a total of 21 modules. Once modules have been selected, the Guide will develop a personalized program for the participant. The participant will then be enrolled into the personalized program. Participants in this group will receive guided support by video chat or phone each week (based on participant's preference) by a trained Guide over the 8-week duration of the program. Weekly contact will include motivating participants to complete the weekly lessons and assistance on the practicing/application of the skills. The Guide will spend approximately 10-15 minutes per week with each participant.
  Interventions: Behavioral: Internet Delivered Cognitive Behavioural Therapy
- Standard ICBT (Active Comparator): Participants in the standard group will receive the ICBT program (containing 21 modules) as is. No personalization will be provided. Similar to the personalized ICBT group, participants will receive guided support by video chat or phone each week (based on participant's preference) by a trained Guide over the 8-week duration of the program. Weekly contact will include motivating participants to complete the weekly lessons and assistance on the practicing/application of the skills. The Guide will spend approximately 10-15 minutes per week with each participant.
  Interventions: Behavioral: Internet Delivered Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Internet Delivered Cognitive Behavioural Therapy — The tinnitus ICBT program consists of 1) an overview of tinnitus, depression, and anxiety; 2) managing unhelpful thoughts and learning problem solving strategies association with pain, anxiety, depression, and disability; 3) management of common symptoms associated with tinnitus, anxiety, and depression; 4) developing strategies to maintain activities while minimizing fatigue; and 5) strategies to improve quality of life through effective goal setting. Supplementary lessons can be accessed at any time (e.g., sleep, communication, problem solving, assertiveness training). Materials are presented in a didactic (i.e., text-based and audio with visual images) and case-enhanced learning format (i.e., stories demonstrate the application of skills). Case vignettes that specifically reflect the experiences of those with tinnitus are included.

SUMMARY:
The goal of this randomized controlled trial is to learn if guided Internet-delivered Cognitive Behavioural Therapy can treat tinnitus-related distress and its associated comorbidities such as anxiety, depression, insomnia, and quality of life among adult tinnitus patients in Canada. The main questions it aims to answer are:

* Does guided internet-delivered cognitive behavioural therapy for the treatment of tinnitus reduce tinnitus-related distress and tinnitus-associated comorbidities (depression, anxiety, insomnia, quality of life) among adult tinnitus patients aged 18-79 years in Canada from pre-treatment to post-treatment and 3-month follow-up?
* Do participants in the personalized ICBT treatment group show worse improvements in patient-reported outcomes from pre-treatment to post-treatment and 3-month follow-up than the standard ICBT control group?

The researchers will compare a personalized ICBT program to a standard ICBT program to investigate if participants in the personalized ICBT program will show no worse improvements in patient-reported outcomes from pre-treatment to post-treatment and 3-month follow-up than the active comparator, the standard ICBT program.

Participants will:

* Receive either a personalized ICBT program or a standard ICBT program delivered over 8 weeks consisting of 21 modules.
* Receive guided support of approximately 10-15 minutes per week by video chat or phone from a trained Guide over the 8-week duration of the program.
* Complete assessments at baseline, post-intervention, and 3-month follow-up through online REDCap surveys with automatic emails and telephone reminders.

DETAILED DESCRIPTION:
Tinnitus is a condition where people hear sounds like ringing or buzzing without an external sound producing source. Tinnitus affects millions globally and is linked to poor mental health, including depression, anxiety, and insomnia. Current treatments have limited success, and Cognitive Behavioral Therapy (CBT) is the most effective, though rarely available.

The study aims to test a personalized, internet-delivered CBT (ICBT) program for tinnitus sufferers in Canada. This program could offer a cost-effective, accessible treatment option. The study will compare a personalized ICBT program with a standard ICBT program to evaluate their effectiveness in reducing tinnitus distress and improving related conditions like depression, anxiety, insomnia and quality of life.

The study will involve 82 participants, who will be randomly assigned to either the personalized or standard ICBT group. Both groups will receive guided support over eight weeks. The research hopes to demonstrate that the personalized ICBT is as effective as the standard ICBT program, but with added benefits in convenience and cost.

ELIGIBILITY:
Inclusion Criteria:

1. adults (18-79 years);
2. diagnosed with tinnitus for more than 6 months;
3. ability to read and write in English;
4. cognitive capacity to consent and participate in the therapeutic process;
5. able to access the technology required for the program (telephone, computer, internet);
6. Canadian residents;
7. A score of 25 or above on the Tinnitus Functional Index (TFI) suggesting the need for tinnitus care.

Exclusion Criteria:

1. have significant cognitive impairments that impact their ability to participate in the therapy;
2. are currently involved in another psychotherapeutic intervention on a regular basis;
3. present with severe mental health disorder that would be better treated in person (e.g., severe suicide ideation, severe substance abuse, recent history of psychosis, mania);
4. have tinnitus as a consequence of a medical disorder, still under investigation;
5. are reporting objective, pulsatile, or unilateral tinnitus, which have not been investigated medically;
6. are undergoing any tinnitus therapy concurrently with partaking in this study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Tinnitus distress | baseline, post-treatment and 3-month follow-up
  The primary assessment measure to quantify distress will be the Tinnitus Functional Index (TFI). A 13-point change in TFI scores will be identified as a clinically meaningful/significant change. Low scores indicate low severity and high scores indicate high severity.

SECONDARY OUTCOMES:
Depression | baseline, post-treatment and 3-month follow-up
  The Patient Health Questionnaire-9 (PHQ-9) will be used to measure depression. Low scores indicate low severity and high scores indicate high severity.
Anxiety | baseline, post-treatment and 3-month follow-up
  Generalized Anxiety Disorder-7 (GAD-7) will be used to measure anxiety. Low scores indicate low severity and high scores indicate high severity.
Insomnia | baseline, post-treatment and 3-month follow-up
  Insomnia Severity Index (ISI) will be used to measure insomnia. Low scores indicate low severity and high scores indicate high severity.
Satisfaction with life | baseline, post-treatment and 3-month follow-up
  Satisfaction with Life Scales (SWLS) for satisfaction with life will be used to measure satisfaction with life. Low scores indicate low satisfaction and high scores indicate high satisfaction.
Hearing Handicap | baseline, post-treatment and 3-month follow-up
  Hearing Handicap Inventory for Adults Screening version (HHIA-S) will be used to measure hearing handicap. Low scores indicate low severity and high scores indicate high severity.
Cost effectiveness | 3-month follow-up
  Productivity Cost Questionnaire (iPCQ) will be used to measure cost-effectiveness.
Healthcare usage | 3-month follow-up
  Medical Consumption Questionnaire (iMCQ) will be used to measure health care usage

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No